CLINICAL TRIAL: NCT01055405
Title: Phase IV Study on the Effects of Sildenafil in Combination With Pulmonary Rehabilitation Program on Exercise Tolerance in Patients With COPD and Pulmonary Hypertension
Brief Title: Study of Sildenafil Effects in Combination With Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Associated Pulmonary Hypertension
Acronym: SIL-COPD-02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Joan Albert Barbera Mir, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JA Barbera
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: Exercise tolerance; COPD; Pulmonary hypertension; Sildenafil
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil plus pulmonary rehabilitation (Experimental)
  Interventions: Drug: Sildenafil
- Placebo plus pulmonary rehabilitation (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 20mg TID orally
  Other Names: Revatio
  Arms: Sildenafil plus pulmonary rehabilitation
Other: Placebo — Placebo TID orally
  Arms: Placebo plus pulmonary rehabilitation

SUMMARY:
Sildenafil is a phosphodiesterase-5 inhibitor that has been approved for the treatment of pulmonary arterial hypertension with orphan drug designation. Sildenafil modulates the nitric oxide (NO) pathway in the vessel wall. Since this pathway is impaired in pulmonary arteries of patients with pulmonary hypertension (PH) associated with chronic obstructive pulmonary disease (COPD), the investigators hypothesized that sildenafil might improve pulmonary hemodynamics and increase exercise tolerance in this condition.

DETAILED DESCRIPTION:
It is a prospective, randomized, double-blind, placebo controlled trial to assess the effect of 3 months treatment with sildenafil (20 mg/8 h), added to a pulmonary rehabilitation program, on exercise tolerance. Subjects: 60 patients (30 by treatment group). Main end-point variable: endurance time in constant work exercise test (CWET). Other measurements: 6 min walk distance, performance in incremental exercise test, physiological and metabolic response at iso-time and iso-load in CWET, dyspnea, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* COPD, FEV1 < 80% ref. and FEV1/FVC < 0.7 post bronchodilator
* Age 40-80 years
* Pulmonary hypertension
* Consent to participate in the study

Exclusion Criteria:

* Pulmonary or extrapulmonary disease that modifies gas exchange or pulmonary hemodynamics
* Recent exacerbation (<4 weeks) (temporally)
* Patients treated with nitrates or CYP3A4 inhibitors (ketoconazole, itraconazole, ritonavir)
* Ischemic optic neuropathy
* Patients treated with phosphodiesterase-5 inhibitors
* Patients with ischemic cardiopathy
* Systemic disease that could modified the results
* Patients unable to practise exercise

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Endurance time | 3 months

SECONDARY OUTCOMES:
6 min walk distance, performance in incremental exercise test, physiological and metabolic response at iso-time and iso-load in CWET, dyspnea, and health-related quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joan Albert Barbera, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Blanco I, Santos S, Gea J, Guell R, Torres F, Gimeno-Santos E, Rodriguez DA, Vilaro J, Gomez B, Roca J, Barbera JA. Sildenafil to improve respiratory rehabilitation outcomes in COPD: a controlled trial. Eur Respir J. 2013 Oct;42(4):982-92. doi: 10.1183/09031936.00176312. Epub 2013 Feb 21. PMID 23429918